CLINICAL TRIAL: NCT06111898
Title: Neuro-biomechanical Aspects Determining the Motor Behavior in Infants With High-risk of Neuromotor Impairments
Brief Title: Neuro-biomechanical Determinants for Motor Behavior in High-risk Infants
Acronym: BAMBI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stephane ARMAND, Professor, University Hospital, Geneva
Other Study IDs: 2023-01113
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Premature Birth; Cerebral Palsy; Neurodevelopmental Disorders; Brain Injuries; Nervous System Diseases
Keywords: Brain Imaging; General Movements; 3D freehand ultrasound; Muscle Morphology; Electromyography
MeSH Terms: conditions — Premature Birth; Cerebral Palsy; Neurodevelopmental Disorders; Brain Injuries; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk infants
  Interventions: Other: No Intervention
- Typically developing infants
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
This project focuses on motor development, muscle growth and muscle activity. Using advanced, instrumented tests such as , the link between muscles and the movement characteristics will be studied. In addition, the evolution of these neuro-biomechanical determinants during the first year of life will be investigated. The examinations are planned for a group of high-risk infants (e.g. premature birth, cases of asphyxia, etc.) compared with a group of infants with typical development.

DETAILED DESCRIPTION:
Background and rationale:

Prematurity and the associated causes of perinatal brain damage, as well as neonatal stroke and birth asphyxia, are major risk factors for neurodevelopmental disorders appearing from birth. In addition, these neuromotor disorders resulting from impaired brain development appear progressively over the course of the first year, affecting early movement and muscle growth. Therefore, early diagnosis and motor therapy are essential to improve long-term neurodevelopmental outcomes. However, in order to provide adequate strategies for these high-risk infants, it is crucial to identify the determinants of potential neuromotor deficits and their consequences on early motor behavior and developmental trajectory during the first year of life. A multimodal tool is needed to reveal the early neuro-biomechanical determinants of motor behavior in infants at high risk of neurodevelopmental disorders.

Objective(s):

* Establishing a comprehensive multimodal tool for the assessment of neuro-biomechanical determinants of motor behavior in the first year of life in high-risk infants for neurodevelopmental impairments, further referred to as "advanced muscle and movement analysis (AMMA)"
* Revealing early neuro-biomechanical determinants in high-risk infants covering the first year of life, including the time points in the neonatal period, at term age, at 3 months of (corrected) age, at 6 months of (corrected) age and at 12 months of (corrected) age, by using the AMMA

Outcome(s):

* Using valid and reliable assessments within the protocol
* Differences in neuro-biomechanical determinants between typically developing infants and high-risk infants at each time point.
* Associations between the neuro-biomechanical determinants of motor behaviour in high-risk infants at each time point
* Changes over time and interaction in the neuro-biomechanical determinants, and comparisons of these evolutions in high-risk infants with typical development.

Methodology

The current study is a national, single center (Geneva University Hospitals), observational study. This observational research will perform both cross-sectional and longitudinal data collection for cohorts of live-born infants.

The study population for this study will include children, i.e., neonates and infants between the age of 35-36 weeks of gestational age to 12 months of (corrected) age. Further, two main groups of children will be included, (a) typically developing (TD) children and (b) children at high-risk for neurodevelopmental impairments. The TD children will be used as a control group.

Procedure

Multiple study visits are planned for longitudinal data collection within the first year of life, i.e. a time of term age, at 3 months, at 6 months and 12 months of age. For the preterms, the investigators also plan to perform an assessment in the neonatal period, i.e. 35-36 weeks of gestation.

The duration of each visit session will be around 90 minutes per participant, providing also time for feeding moments and adaptation of the infant to the new environment. The visit in the neonatal period will be organized at the Neonatology Unit at HUG (Geneva University Hospitals). All visits from the term (equivalent) age will be organized in the Kinesiology Laboratory at the HUG.

In general, clinical data such as birth information, structural brain MRI and developmental assessments will be derived from the medical records.

The main procedures during each research visit are:

1. Muscle assessment: using 3D freehand ultrasound technique, measuring the lower legs muscles, assessing muscle volume and length.
2. Neuromotor development: using standardized scales, measuring the gross motor development and motor repertoire, assessing age-appropriate neuromotor development.
3. Motor behavior: using surface electromyography and motion capture system, measuring spontaneous movements, assessing the movement quality and quantity

ELIGIBILITY:
Inclusion & exclusion criteria for group of high-risk infants:

* Infants born before or at 28 weeks of gestation
* Infants born after 28 weeks of gestation and with brain injury.
* A term birth with the clinical diagnosis of asphyxia (ischemic event with hypothermia) or neonatal stroke
* Exclusion in case of genetic syndrome, or lower limb pathology (e.g. spina bifida)

Inclusion & exclusion criteria for group of typically developing children:

* Born at a gestational age above 37 weeks
* Birth weight between P10 and P90
* Head circumference between P10 and P90
* Ph >7.1
* Exclusion in case of genetic syndrome, lower limb pathology and/or brain malformations

Ages: 35 Weeks to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm or a term born Infants with detectable risk factors for neurodevelopmental impairments will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 348 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
General Movement Assessment | 35-36 weeks of gestation; term equivalent age, 3 months (corrected) age
  Observation of general movements following the Prechtl's General Movement Assessment, interpreted by observing age-specific general movement components and extracting the Motor Optimality Score (0-12, the higher, the better outcome)
Hammersmith Neonatal/Infant Neurological Examination | 35-36 weeks of gestation; term equivalent age, 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  Neurological assessment for different domains such as muscle tone, postures, movements and reflexes . Resulting in total scores (0-78) which can be compared to norm values, and higher scores indicate better outcome.
Change in muscle morphology size | 35-36 weeks of gestation; term equivalent age, 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  The size of the lower leg muscles defined by freehand ultrasound
Change in muscle morphology length | 35-36 weeks of gestation; term equivalent age, 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  The length of the lower leg muscles defined by freehand ultrasound
Change in muscle activity | 35-36 weeks of gestation; term equivalent age, 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  Investigation of the muscle activity during spontaneous, whole body movements by using surface electromyography.
Change in motor behaviour | 35-36 weeks of gestation; term equivalent age, 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  Investigation movement quality/quantify during spontaneous, whole body movements by using reflective markers.

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development - Version III | 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  Standardized neurodevelopmental test of gross and fine motor skills. Higher scores indicate better outcome.
Alberta Infant Motor Scale (AIMS) | 3 months (corrected) age, 6 months (corrected) age and 12 months (corrected) age.
  Assessment of gross motor development during prone, supine, sitting and standing. Scores from 0-60. Higher scores indicate better outcome.
Magnetic resonance imaging of the brain: classification | up to 4 weeks post-term age
  Qualitatively assessment on the MRI classification system by Himmelman et al. to classify the nature of brain abnormalities.
Magnetic resonance imaging of the brain: quantification | up to 4 weeks post-term age
  Qualitatively assessment on the MRI classification system by quantitative assessment using the Kidokoro scoring system to classify the extent of white and grey matter abnormalities. Total global scores were classified as normal (0-3), mild (4-7), moderate (8-11), or severe (≥12) brain abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available upon publication via online repository (yareta or zenodo)
Time Frame: Upon publication

REFERENCES:
- [Background] Pascal A, Govaert P, Oostra A, Naulaers G, Ortibus E, Van den Broeck C. Neurodevelopmental outcome in very preterm and very-low-birthweight infants born over the past decade: a meta-analytic review. Dev Med Child Neurol. 2018 Apr;60(4):342-355. doi: 10.1111/dmcn.13675. Epub 2018 Jan 19. PMID 29350401
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Gough M, Shortland AP. Could muscle deformity in children with spastic cerebral palsy be related to an impairment of muscle growth and altered adaptation? Dev Med Child Neurol. 2012 Jun;54(6):495-9. doi: 10.1111/j.1469-8749.2012.04229.x. Epub 2012 Feb 27. PMID 22364585
- [Background] De Beukelaer N, Vandekerckhove I, Huyghe E, Molenberghs G, Peeters N, Hanssen B, Ortibus E, Van Campenhout A, Desloovere K. Morphological Medial Gastrocnemius Muscle Growth in Ambulant Children with Spastic Cerebral Palsy: A Prospective Longitudinal Study. J Clin Med. 2023 Feb 16;12(4):1564. doi: 10.3390/jcm12041564. PMID 36836099
- [Background] Willerslev-Olsen M, Choe Lund M, Lorentzen J, Barber L, Kofoed-Hansen M, Nielsen JB. Impaired muscle growth precedes development of increased stiffness of the triceps surae musculotendinous unit in children with cerebral palsy. Dev Med Child Neurol. 2018 Jul;60(7):672-679. doi: 10.1111/dmcn.13729. Epub 2018 Mar 24. PMID 29573407
- See also: Grant description — https://data.snf.ch/grants/grant/212517